CLINICAL TRIAL: NCT05158335
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of Single and Multiple Ascending Doses of MBX 2109 in Healthy Participants
Brief Title: Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of MBX 2109 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MBX Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: MBX-2H1001
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MBX 2109 (Part A) (Experimental): Single ascending SC doses
  Interventions: Drug: MBX 2109 (Part A)
- MBX 2109 (Part B) (Experimental): Repeated ascending SC doses
  Interventions: Drug: MBX 2109 (Part B)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBX 2109 (Part A) — Single ascending SC dose of MBX 2109: 50 µg, 150 µg, 300 µg, 460 µg, 600 µg
  Arms: MBX 2109 (Part A)
Drug: MBX 2109 (Part B) — Repeated ascending SC doses of MBX 2109: 200 µg, 300 µg, 460 µg, 600 µg, 900 µg
  Arms: MBX 2109 (Part B)
Drug: Placebo — Single SC dose or repeated SC doses of placebo.
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple doses of MBX 2109 in healthy volunteers.

This study includes 2 parts. Part A involves a single dose of MBX 2109 taken as a subcutaneous (SC) injection just under the skin. Part B involves repeat doses of MBX 2109 taken as a SC injection just under the skin. Each participant will enroll in only one part.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women (of nonchildbearing potential) between 20 and 60 years of age, inclusive.
2. Body mass index between 20.0 and 32.0 kg/m2, inclusive.
3. No clinically meaningful findings on physical examination, electrocardiogram, laboratory tests or vital signs
4. Subject has been given signed informed consent

Exclusion Criteria:

1. History of any significant illness or disorder
2. Acute illness within 30 days of administration of first dose of study drug
3. Positive screening result for HIV, hepatitis B or hepatitis C
4. History of or current substance abuse (drug or alcohol) within past 1 year or positive test for drugs of abuse during screening
5. Use of nicotine-containing or vaping products within 3 months prior to screening or check-in
6. Use of cannabis within 45 days prior to check-in
7. Donation of blood within 3 months prior to screening, plasma within 2 weeks prior to screening or platelets within 6 weeks prior to screening
8. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within past 30 days

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men and women of non-child bearing potential
Enrollment: 76 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures | Baseline through Day 40 (part A) or Day 60 (Part B)
  Number of participants with adverse events (AEs) or Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Secondary Outcome Measures 1 | Baseline through Day 40 (part A) or Day 60 (Part B)
  Pharmacokinetics (PK): Area Under the Concentration versus Time Curve (AUC) of MBX 2109
Secondary Outcome Measures 2 | Baseline through Day 40 (part A) or Day 60 (Part B)
  Pharmacodynamics (PD): change from baseline in albumin corrected serum calcium

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Geiger, MD, PhD, Study Director — MBX Biosciences
Locations (2):
- United States (2):
  - Labcorp Drug Development: Clinical Research Unit, Dallas, Texas
  - Labcorp Drug Development: Clinical Research Unit, Madison, Wisconsin